CLINICAL TRIAL: NCT07289776
Title: A Randomized, Single-center, Double-blind, Placebo-controlled, First-in-human Trial With Single and Multiple Ascending Doses to Determine Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GRT7041 in Healthy Participants.
Brief Title: A First-in-human Trial of GRT7041 in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP7041-01
Record Dates: First submitted 2025-11-24; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Treatment of Pain
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1: SAD (Experimental): With up to five cohorts SAD1 to SAD5 (n = 40). To be conducted in adult males and WONCBP
  Interventions: Drug: GRT7041 SAD; Drug: Placebo
- Part 2: MAD (Experimental): With up to three cohorts, MAD1 to MAD3 (n = 30) dosed once daily (QD) for a period of 14 days. To be conducted in adult males only.
  Interventions: Drug: Placebo; Drug: Midazolam; Drug: GRT7041 MAD

INTERVENTIONS:
Drug: GRT7041 SAD — Single ascending doses
  Arms: Part 1: SAD
Drug: Placebo — Placebo to match GRT7041 dose strength
Drug: Midazolam — Solution
  Arms: Part 2: MAD
Drug: GRT7041 MAD — Multiple ascending doses
  Arms: Part 2: MAD

SUMMARY:
The purpose of this trial is to assess the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of GRT7041 in healthy male and female (Women of non-childbearing potential) participants.

The trial duration will be up to approximately 6 weeks for participants in Part 1 (Single ascending dose [SAD]), except for participants taking part in the food effect cohort SAD3 where the trial duration will be up to approximately 8 weeks. The trial duration will be up to approximately 7 weeks in Part 2 (Multiple ascending dose [MAD]), and the Treatment Period will be up to 14 days (for Part 2).

The trial will include a Screening Visit, an in-house stay period and Follow-up (FU) Visit/End-of-Trial (EoT) Visit.

DETAILED DESCRIPTION:
The trial will consist of two parts:

* Part 1: SAD with up to five cohorts SAD1 to SAD5 (n = 40). To be conducted in adult males and women of non-childbearing potential (WONCBP).
* Part 2: MAD with up to three cohorts, MAD1 to MAD3 (n = 30) dosed once daily (QD) for a period of 14 days. To be conducted in adult males only.

The trial design also evaluate the potential interaction of GRT7041 with a CYP3A4 index substrate that will be assessed separately in all cohorts in Part 2 (MAD) of the trial.

Dosing in Parts 1 and 2 will be conducted under fasted conditions, except for the SAD3 cohort in Part 1 (SAD), where participants will also receive a standardized breakfast (SAD3b treatment) to assess the effect of food.

ELIGIBILITY:
Main Inclusion Criteria:

1. The participant must be able to give signed informed consent, including compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Participants must sign the ICF before any trial-related assessments.
3. The participant is in good health as judged by the Investigator including medical history, physical examination, 12-lead ECG, vital signs (pulse rate, respiratory rate, systolic and diastolic BP), body temperature, and clinical laboratory parameters (clinical chemistry, hematology, coagulation and urinalysis) without clinically relevant deviations from reference ranges, unless further specified in the exclusion criteria.

Main Exclusion Criteria:

1. History of any of the following: cardiac impairment, renal impairment, pancreatitis, coagulation abnormalities.
2. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk for treatment complications/ participation in the trial unsafe.
3. Any disease or conditions known to interfere with the absorption, distribution, metabolism, or excretion of the IMP.
4. Evidence or medical history of clinically significant and relevant psychiatric issues as assessed by the Investigator.
5. Confirmed or suspected history of clinically relevant drug allergy.
6. Major surgical procedure, within 30 days prior to ICF signing, or anticipation of need for a major surgical procedure during the trial.
7. Blood loss of 500 mL or more (eg, owing to blood donation) within 90 days before Screening Visit.
8. The participant has used any medication, including herbal remedies or over-the-counter medication within 2 weeks (or 5 half-lives, whichever is longer) before the start of the trial intervention or anticipated use during the trial, unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the trial.
9. The participant is enrolled in another clinical trial unless it is an observational (non-interventional) clinical trial or during the follow-up period of an interventional trial) or has received an IMP in another clinical trial within 30 days before Day 1 or within 5 times the elimination half-life of the IMP, whichever is longer.
10. Reluctance to comply with contraception requirements.
11. Evidence or history of alcohol or drug abuse including positive or missing alcohol breath test or drugs of abuse test(s).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The participant is biologically male (both Part 1 and Part 2) or biological female of non-childbearing potential (Part 1 only).
Enrollment: 70 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2026-08-24 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | Through study completion, an average of 8 Weeks
  An AE is defined as any unfavorable medical occurrence in a trial participant administered the investigational product.
  Assessment of the safety and tolerability of GRT7041 after oral single and multiple-dose escalation
Number of participants with Serious Adverse Events | Through study completion, an average of 8 Weeks
  A Serious Adverse Event (SAE) is any untoward medical occurrence that, at any dose:
  * Results in death, is life-threatening, or requires (or prolongs) hospitalization;
  * Results in persistent or significant disability/incapacity;
  * Is a congenital anomaly or birth defect; or
  * Is considered medically significant, requiring intervention to prevent one of the outcomes above.
  * Investigator judgment applies to other clinically important events that may not be immediately life-threatening but could jeopardize participant safety.
  Assessment of the safety and tolerability of GRT7041 after oral single and multiple-dose escalation

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve from 0 to 24 hours [(AUC)0-24] [SAD] | Day 1 to Day 4 (Pre-dose, 0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 18 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours) and Day 10 (240 hours)
  The total amount of the study drug (and metabolite) in the blood during the first 24 hours after it is taken.
  Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Area Under the Plasma Concentration-Time Curve from Time 0 to the last measurable concentration (t) [AUC0-t] [SAD] | Day 1 to Day 4 (Pre-dose, 0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 18 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours) and Day 10 (240 hours)
  The total amount of the study drug (and metabolite) in the blood from the time it is taken until the last time a measurable level of the drug is found.
  Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Area Under the Plasma Concentration-Time Curve from Time 0 extrapolated to infinity (AUC0-inf ) [SAD] | Day 1 to Day 4 (Pre-dose, 0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 18 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours) and Day 10 (240 hours)
  The total amount of the study drug (and metabolite) in the blood from the time it is taken until it has completely left the body.
  Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Maximum Observed Plasma Concentration (Cmax) [SAD] | Day 1 to Day 4 (Pre-dose, 0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 18 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours) and Day 10 (240 hours)
  The maximum amount of the study drug (and metabolite) measured in the blood after taking the dose.
  Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Time to Reach Maximum Observed Plasma Concentration (Tmax) [SAD] | Day 1 to Day 4 (Pre-dose, 0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 18 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours) and Day 10 (240 hours)
  The time it takes to reach the highest concentration of the study drug (and metabolite) in the blood after dosing.
  Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Terminal Elimination Half-Life (t₁/₂) [SAD] | Day 1 to Day 4 (Pre-dose, 0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 18 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours) and Day 10 (240 hours)
  The time it takes for the amount of study drug (and metabolite) in the blood to reduce by half after reaching its peak level.
  Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Terminal Elimination Rate Constant (λz) [SAD] | Day 1 to Day 4 (Pre-dose, 0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 18 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours) and Day 10 (240 hours)
  The rate at which the study drug (and metabolite) is eliminated from the blood during the final phase after dosing.
  Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Apparent Total Clearance of Drug From Plasma After Extravascular Administration (CL/F) [SAD] | Day 1 to Day 4 (Pre-dose, 0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 18 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours) and Day 10 (240 hours)
  The amount of blood completely cleared of thestudy drug (and metabolite) per unit of time, taking into account how much of the drug is absorbed into the body.
  Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Apparent Volume of Distribution During the Terminal Phase After Extravascular Administration (Vz/F) [SAD] | Day 1 to Day 4 (Pre-dose, 0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 18 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours) and Day 10 (240 hours)
  An estimate of how widely the study drug spreads through the body's tissues after it is absorbed.
  Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Lag Time Before First Measurable Concentration (tlag) [SAD] | Day 1 to Day 4 (Pre-dose, 0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 18 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours) and Day 10 (240 hours)
  The time between when the study drug (and metabolite) is taken and when it first becomes measurable in the blood.
  Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Time of Last Measurable Concentration (tlast) [SAD] | Day 1 to Day 4 (Pre-dose, 0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 18 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours) and Day 10 (240 hours)
  The last time point when a measurable amount of the study drug (and metabolite) is found in the blood.
  Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Amount of Study Drug Excreted in Urine (Ae) [SAD] | Day 1 to Day 4 (from 0 hours to 72 hours)
  The total amount of the study drug (and metabolite) that is passed out of the body through urine during a specific collection period.
  Collected only for one cohort in Part 1: SAD.
  Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Cumulative Amount of Study Drug Excreted in Urine (Cumulative Ae) [SAD] | Day 1 to Day 4 (from 0 hours to 72 hours)
  The total amount of the study drug (and metabolite) eliminated in urine from the time of dosing up to the end of each collection period, showing how much of the drug has been removed from the body over time.
  Collected only for one cohort in Part 1: SAD. Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Percentage of Dose Excreted in Urine (Ae%) [SAD]. | Day 1 to Day 4 (from 0 hours to 72 hours)
  The percentage of the total amount of the study drug (and metabolite) dose that is passed out in urine during each collection period.
  Collected only for one cohort in Part 1: SAD. Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Cumulative Percentage of Dose Excreted in Urine (Cumulative Ae%) [SAD] | Day 1 to Day 4 (from 0 hours to 72 hours)
  The total percentage of the study drug dose excreted in urine from dosing until the end of each collection period, showing how much of the drug has been eliminated over time.
  Collected only for one cohort in Part 1: SAD. Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Renal Clearance of Study Drug (CLr) [SAD] | Day 1 to Day 4 (from 0 hours to 72 hours)
  The rate at which the study drug (and metabolite) is removed from the blood by the kidneys and excreted in the urine.
  Collected only for one cohort in Part 1: SAD. Assessment of the PK of GRT7041 and its metabolite, GRT1093025, for single-dosing.
Area Under the Concentration-Time Curve from 0 to 24 hours [(AUC)0-24] [MAD] | Day 1 (0 hours - 24 hours)
  Assessment of the pharmacokinetics (PK) of GRT7041 and its metabolite, GRT1093025, for multiple-dosing.
Maximum Observed Plasma Concentration (Cmax) [MAD] | Day 1 (0 hours - 24 hours)
  Assessment of the pharmacokinetics (PK) of GRT7041 and its metabolite, GRT1093025, for multiple-dosing.
Time to Reach Maximum Observed Plasma Concentration (Tmax) [MAD] | Day 1 (0 hours - 24 hours)
  Assessment of the pharmacokinetics (PK) of GRT7041 and its metabolite, GRT1093025, for multiple-dosing.
Area Under the Plasma Concentration-time Curve Over a Dose Interval at Steady State (AUCτ,ss) [MAD] | Day 14 - Day 17 (0 hours to 72 hours after last dose) and Day 21
  Assessment of the pharmacokinetics (PK) of GRT7041 and its metabolite, GRT1093025, for multiple-dosing
Maximum Observed Plasma Concentration at Steady State (Cmax,ss) [MAD] | Day 14 - Day 17 (0 hours to 72 hours after last dose) and Day 21
  Assessment of the pharmacokinetics (PK) of GRT7041 and its metabolite, GRT1093025, for multiple-dosing
Minimum Observed Plasma Concentration at Steady State (Cmin,ss) [MAD] | Day 1, Day 2, Day 4, Day 6, Day 8, Day 10, and Day 12 to Day 17 and Day 21
  Assessment of the pharmacokinetics (PK) of GRT7041 and its metabolite, GRT1093025, for multiple-dosing
Average Observed Plasma Concentration at Steady State (Cav.ss) [MAD] | Day 1, Day 2, Day 4, Day 6, Day 8, Day 10, and Day 12 to Day 17 and Day 21
  Assessment of the pharmacokinetics (PK) of GRT7041 and its metabolite, GRT1093025, for multiple-dosing
Time to Reach Maximum Observed Plasma Concentration (Tmax) at Steady State (tmax,ss) [MAD] | Day 14 - Day 17 (0 hours to 72 hours after last dose) and Day 21
  Assessment of the pharmacokinetics (PK) of GRT7041 and its metabolite, GRT1093025, for multiple-dosing
Terminal Elimination Half-Life (t₁/₂) [MAD] | Day 1, Day 2, Day 4, Day 6, Day 8, Day 10, and Day 12 to Day 17 and Day 21
  Assessment of the pharmacokinetics (PK) of GRT7041 and its metabolite, GRT1093025, for multiple-dosing
Terminal Elimination Rate Constant (λz) [MAD] | Day 1, Day 2, Day 4, Day 6, Day 8, Day 10, and Day 12 to Day 17 and Day 21
  Assessment of the pharmacokinetics (PK) of GRT7041 and its metabolite, GRT1093025, for multiple-dosing
Apparent Total Clearance of Drug From Plasma After Extravascular Administration (CL/F) [MAD] | Day 1, Day 2, Day 4, Day 6, Day 8, Day 10, and Day 12 to Day 17 and Day 21
  Assessment of the pharmacokinetics (PK) of GRT7041 and its metabolite, GRT1093025, for multiple-dosing
Apparent Volume of Distribution During the Terminal Phase After Extravascular Administration (Vz/F) [MAD] | Day 1, Day 2, Day 4, Day 6, Day 8, Day 10, and Day 12 to Day 17 and Day 21
  Assessment of the pharmacokinetics (PK) of GRT7041 and its metabolite, GRT1093025, for multiple-dosing
Time of Last Measurable Concentration (tlast) [MAD] | Day 14 - Day 17 (0 hours to 72 hours after last dose) and Day 21
  Assessment of the pharmacokinetics (PK) of GRT7041 and its metabolite, GRT1093025, for multiple-dosing
Maximum Observed Plasma Concentration (Cmax) [SAD] for fed and fasted state | Day 1 to Day 4 (Pre-dose, 0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 18 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours) and Day 10 (240 hours)
  Assessment of the effect of food on the PK of GRT7041 following single-dosing
Area Under the Plasma Concentration-Time Curve from Time 0 to the last measurable concentration (t) [AUC0-t] [SAD] for fed and fasted state | Day 1 to Day 4 (Pre-dose, 0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 18 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours) and Day 10 (240 hours)
  Assessment of the effect of food on the PK of GRT7041 following single-dosing
Area Under the Plasma Concentration-Time Curve from Time 0 extrapolated to infinity (AUC0-inf ) [SAD] for fed and fasted state | Day 1 to Day 4 (Pre-dose, 0 minutes, 15 minutes, 30 minutes, 45 minutes, 1 hour 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours, 18 hours, 24 hours, 30 hours, 36 hours, 48 hours, 72 hours) and Day 10 (240 hours)
  Assessment of the effect of food on the PK of GRT7041 following single-dosing
Area Under the Plasma Concentration-Time Curve from Time 0 to the last measurable concentration (t) [AUC0-t] of midazolam | Day -1, Day 1 and Day 14 (pre-dose, 0.25 hours, 0.5 hours, 1 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours and 18 hours)
  PK parameters (AUC0-t, AUC0-inf, Cmax, tmax and t1/2) of midazolam (index substrate) before and after treatment with GRT7041 over 14 days, and when administered alone and after single day and 14 days of treatment with GRT7041
Area Under the Plasma Concentration-Time Curve from Time 0 extrapolated to infinity (AUC0-inf ) of midazolam | Day -1, Day 1 and Day 14 (pre-dose, 0.25 hours, 0.5 hours, 1 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours and 18 hours)
  PK parameters (AUC0-t, AUC0-inf, Cmax, tmax and t1/2) of midazolam (index substrate) before and after treatment with GRT7041 over 14 days, and when administered alone and after single day and 14 days of treatment with GRT7041
Maximum Observed Plasma Concentration (Cmax) of midazolam | Day -1, Day 1 and Day 14 (pre-dose, 0.25 hours, 0.5 hours, 1 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours and 18 hours)
  PK parameters (AUC0-t, AUC0-inf, Cmax, tmax and t1/2) of midazolam (index substrate) before and after treatment with GRT7041 over 14 days, and when administered alone and after single day and 14 days of treatment with GRT7041
Time to Reach Maximum Observed Plasma Concentration (Tmax) of midazolam | Day -1, Day 1 and Day 14 (pre-dose, 0.25 hours, 0.5 hours, 1 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours and 18 hours)
  PK parameters (AUC0-t, AUC0-inf, Cmax, tmax and t1/2) of midazolam (index substrate) before and after treatment with GRT7041 over 14 days
Terminal Elimination Half-Life (t₁/₂) of midazolam | Day -1, Day 1 and Day 14 (pre-dose, 0.25 hours, 0.5 hours, 1 hours, 1.5 hours, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 10 hours, 12 hours, 15 hours and 18 hours)
  PK parameters (AUC0-t, AUC0-inf, Cmax, tmax and t1/2) of midazolam (index substrate) before and after treatment with GRT7041 over 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- New Zealand Clinical Research (NZCR), Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Group Web Site (see URL below for details); according to the European Federation of Pharmaceutical Industries and Associations (EFPIA) Data Sharing Principles.
URL: https://www.grunenthal.com/en/science/clinical-trials/data-sharing-clinical-trials